CLINICAL TRIAL: NCT05003375
Title: Physiological Responses in Experimentally Induced Cognitive Fatigue in People With Multiple Sclerosis (MS): a Feasibility Study
Brief Title: Physiological Responses in Experimentally Induced Cognitive Fatigue in People With Multiple Sclerosis (MS)
Acronym: PREFIMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Daphne Kos, Associate Professor, KU Leuven
Other Study IDs: S63552
Record Dates: First submitted 2021-01-25; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis; Fatigue; Stress
Keywords: fatigability; cognitive fatigue; cognitive fatigability
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis (MS): People with MS diagnosis, aged 18-55 years, Relapsing Remitting type, EDSS < 6.0, normal vision (if necessary corrected), Dutch speaking.
  Interventions: Behavioral: High-challenging cognitive protocol to provoke stress and (cognitive) fatigue
- Healthy Controls (HC): Healthy controls without relevant health conditions (diabetes, thyroid diseases, neurological disorders), non-pregnant, aged 18-55 years, normal vision (if necessary corrected), Dutch speaking.
  Interventions: Behavioral: High-challenging cognitive protocol to provoke stress and (cognitive) fatigue

INTERVENTIONS:
Behavioral: High-challenging cognitive protocol to provoke stress and (cognitive) fatigue — Baseline measurement is done in two parts: 1) resting for five minutes (no talking, no movement) and 2) speaking at normal pace (2 minutes).
  This is immediately followed by a measurement of the physiological response variables during the testing, in which the following protocol is performed in the order presented: 1) SDMT-NBack task-SDMT*-NBacktask**, 2) NBack task-SDMT-NBack task-SDMT. Participants will run either sequence to check for effects of the previous testing. During the conduct of the study, it will be ensured that half of the participants in each group followed Sequence 1 and the other half of the group followed Sequence 2.
  During all these measurements, the participant will sit at a table with a computer on which the tests are performed.
  *SDMT: Symbol Digit Modalities Test: see description in outcome measures
  **N-Back Task: see description in outcome measures

SUMMARY:
The current study will add to the current knowledge by combining several electrophysiological techniques to examine the relationship between physiological responses and cognitive fatigue and daily activity performance in a stress- and fatigue-inducing protocol.

The aims of this study are: 1) to evaluate the feasibility and usability of assessing physiological responses in an experimental set-up and 2) to investigate the association between physiological outcomes, experimentally induced stress and cognitive fatigue in people with multiple sclerosis (MS) and healthy controls.

DETAILED DESCRIPTION:
In an experimental set-up participants (20 people with MS and 20 healthy controls) will perform a high-challenging cognitive protocol to provoke stress and (cognitive) fatigue.

Physiological responses (heart rate variability, skin conductance, body temperature) and brain activity (EEG) will be measured while resting (resting baseline), while speaking as normal (speaking baseline), during protocol performance and following the protocol (post-protocol).

Demographic and clinical characteristics, as well as levels of perceived fatigue, stress, pain, daily activity performance, quality of life and anxiety and depression will be assessed using medical records and questionnaires.

Feasibility and usability will be assessed in participants and researcher(s) by standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis MS, Relapsing Remitting (RR) type (MS group)
* Expanded Disability Status Scale (EDSS) <6 (MS group)
* Dutch speaking
* normal or corrected vision
* feasible use of computer

Exclusion Criteria:

* relapse < 3 months (MS group)
* pregnancy
* relevant comorbidity (thyroid disease, diabetes, other neurological disorders, metabolic diseases, neuro-endocrine tumor(s)
* severe cognitive disability

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A convenience sample of 20 people with currently stable multiple sclerosis (MS) between 18 and 55 years old and able to walk for 100m will be recruited from the National MS Center Melsbroek, as well as 20 age-matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability (time-domain) | immediately post protocol (approx. 2 hours after baseline)
  ECG monitoring will be done using the MindMedia NEXUS-10MKII.- Heart Rate Variability will be studied in a time- and frequency domain. For the time-domain following measures are studied: 1) the average normal-normal interval; 2) the standard deviation of normal-normal (SDNN); 3) the Root Mean Square of Successive Differences (RMSSD); 4) the percentage of adjacent normal-normal intervals with differences of more than 50miliseconds. (PNN50).
Change in heart rate variability (frequency-domain) | immediately post protocol (approx. 2 hours after baseline)
  ECG monitoring will be done using the MindMedia NEXUS-10MKII.- Heart Rate Variability will be studied in a time- and frequency domain. For the frequency domain, the changes in the high frequency (HF) and low frequency (LF) will be studied and analysed.

SECONDARY OUTCOMES:
Change in Visual Analogue Scale (VAS) Momentary fatigue | immediately post protocol (approx. 2 hours after baseline)
  Momentary fatigue experienced following the protocol using Visual Analogue Scale (VAS) (minimum 0- maximum 10), higher scores indicate higher fatigue.
Change in Visual Analogue Scale (VAS) Momentary pain | immediately post protocol (approx. 2 hours after baseline)
  Momentary pain experienced following the protocol using Visual Analogue Scale (minimum 0- maximum 10), higher scores indicate higher pain.
Usefulness, Satisfaction, and ease of use Questionnaire (USE) | post protocol (approx. 2 hours after baseline)
  The USE is a self-report questionnaire in which 30 items in four dimensions (usefulness, ease of use, ease of learning and satisfaction) are answered on a 7-point Likert scale (1 = disagree, 7 = fully agree) and one not -answer option.
  Higher scores indicate higher satisfaction and usefulness.
NASA Task Load Index (NASA-TLX) | post protocol (approx. 2 hours after baseline)
  The NASA-TLX is a self-report questionnaire that measures perceived work-related stress using six dimensions with a focus on mental stress: mental, physical and time-related stress, frustration and execution. The dimensions are assessed on the basis of a semantic differential scale (0-10). The six individual scores are converted to a global score by means of a "paired comparison task" in which "comparison cards" are used prior to the assessment.
  Higher scores indicate higher task load.
Galvanic Skin Response (GSR) | baseline
  * For the monitoring of the GSR, the Mind Media NEXUS-10MKII will be used.
  * Two electrodes will be placed on the palmar side of the left manus. The first electrode is positioned on the phalanx medialis of the index, the second electrode is positioned on the phalanx medialis of the digitus annulare.
  * As the participants will not be exposed to abrupt changes in stimulus presentation, and no expected or unexpected changes in the environment will be present, the tonic Skin Conductance Level (SCL) will be analysed.
Galvanic Skin Response (GSR) | during protocol (approx. 1 hour after baseline)
  * For the monitoring of the GSR, the Mind Media NEXUS-10MKII will be used.
  * Two electrodes will be placed on the palmar side of the left manus. The first electrode is positioned on the phalanx medialis of the index, the second electrode is positioned on the phalanx medialis of the digitus annulare.
  * As the participants will not be exposed to abrupt changes in stimulus presentation, and no expected or unexpected changes in the environment will be present, the tonic Skin Conductance Level (SCL) will be analysed, using mean microsiemens.
Galvanic Skin Response (GSR) | immediately post protocol (approx. 2 hours after baseline)
  * For the monitoring of the GSR, the Mind Media NEXUS-10MKII will be used.
  * Two electrodes will be placed on the palmar side of the left manus. The first electrode is positioned on the phalanx medialis of the index, the second electrode is positioned on the phalanx medialis of the digitus annulare.
  * As the participants will not be exposed to abrupt changes in stimulus presentation, and no expected or unexpected changes in the environment will be present, the tonic Skin Conductance Level (SCL) will be analysed, using mean microsiemens.
Brain activity | baseline
  • Electroencephalography (EEG):
  * EEG monitoring will be done using the MindMedia NEXUS-10MKII.
  * Ten20 conductive paste for EEG is used in combination with Ag/AgCl disc electrodes.
  * A positive electrode will be placed on Cz according to the international 10-20 system, a negative electrode will be placed on the left earlobe, and the ground electrode for EEG and ECG measurement will be placed on the right earlobe.
  EEG measures:
  - The impact of the cognitive fatigue and stress inducing protocol on alpha, beta, delta, and there frequency bands will be studied.
Brain activity | during protocol (approx. 1 hour after baseline)
  • Electroencephalography (EEG):
  * EEG monitoring will be done using the MindMedia NEXUS-10MKII.
  * Ten20 conductive paste for EEG is used in combination with Ag/AgCl disc electrodes.
  * A positive electrode will be placed on Cz according to the international 10-20 system, a negative electrode will be placed on the left earlobe, and the ground electrode for EEG and ECG measurement will be placed on the right earlobe.
  EEG measures:
  - The impact of the cognitive fatigue and stress inducing protocol on alpha, beta, delta, and there frequency bands will be studied.
Brain activity | immediately post protocol (approx. 2 hours after baseline)
  • Electroencephalography (EEG):
  * EEG monitoring will be done using the MindMedia NEXUS-10MKII.
  * Ten20 conductive paste for EEG is used in combination with Ag/AgCl disc electrodes.
  * A positive electrode will be placed on Cz according to the international 10-20 system, a negative electrode will be placed on the left earlobe, and the ground electrode for EEG and ECG measurement will be placed on the right earlobe.
  EEG measures:
  - The impact of the cognitive fatigue and stress inducing protocol on alpha, beta, delta, and there frequency bands will be studied.
Respiration | baseline
  Respiration set up:
  * The mind media NEXUS-10 MKII will be used for respiration measurement.
  * An elastic band with sensor will be worn around the trunk at height of the umbilicus.
  Respiration measures:
  * Data will solely cover mechanical aspects of breathing.
  * Only the respiration rate will be taken into analyses to study relations with previous neurophysiological measures.
  * Also the breathing rate (BRPM) per minute will be analysed.
Respiration | during protocol (approx. 1 hour after baseline)
  Respiration set up:
  * The mind media NEXUS-10 MKII will be used for respiration measurement.
  * An elastic band with sensor will be worn around the trunk at height of the umbilicus.
  Respiration measures:
  * Data will solely cover mechanical aspects of breathing.
  * Only the respiration rate will be taken into analyses to study relations with previous neurophysiological measures.
  * Also the breathing rate (BRPM) per minute will be analysed.
Respiration | immediately post protocol (approx. 2 hours after baseline)
  Respiration set up:
  * The mind media NEXUS-10 MKII will be used for respiration measurement.
  * An elastic band with sensor will be worn around the trunk at height of the umbilicus.
  Respiration measures:
  * Data will solely cover mechanical aspects of breathing.
  * Only the respiration rate will be taken into analyses to study relations with previous neurophysiological measures.
  * Also the breathing rate (BRPM) per minute will be analysed.
Decline in Symbol Digit Modalities Test | immediately post protocol (approx. 2 hours after baseline)
  The Symbol Digit Modalities Test (SDMT) Performance
  * The SDMT is frequently used in the normal treatment and follow up of people with MS. Therefore, a customized version for this study is developed.
  * Participants are shown one file with at the top a row as example consisting of symbols with related numbers. Beneath this row, a couple of rows with symbols are shown. The participant has to link the number to the specific symbol according to the example row. This as fast as possible within 90 seconds.
  Scores
  * A total score consisting of the total amount of correct answers will be determined.
  * The SDMT will be divided in three equal parts of 30 seconds.
  * For part1 part2, and part3 a correct score will be determined.
  * Additionally, a cognitive fatigability score is determined: the difference between part3 versus part1.
Decline in N-Back Task | immediately post protocol (approx. 2 hours after baseline)
  The N-Back Task (NBT)
  Performance:
  * The participants are shown a presentation of a series of letters. The participants have to respond with 'yes' whenever the same letter appeared as two letters previously.
  * The participants perform two versions of this: with a 2- and 1-second interstimulus interval.
  Scores:
  * A total score consisting of the total amount of correct answers is determined.
  * The NBT is then divided in three equal parts. For part1, part2, and part3, a total correct score is determined.
  * Additionally, a cognitive fatigability score (i.e. difference between part3 and part1) is determined.

OTHER OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | baseline
  The MFIS is a self-report questionnaire used to measure the perceived impact of fatigue on physical, cognitive and psychosocial functioning. The participant answers 21 items on the basis of a 5-point Likert scale (0 = never; 5 = almost always). A higher score on the subscales (physical dimension: 0-36; cognitive dimension: 0-40; psychosocial functioning: 0-8) or in the total score represents a higher degree of fatigue.
Perceived Stress Scale (PSS) | baseline
  Questionnaire on perceived stress in daily life (14 items) The Perceived Stress Scale (PSS) is a self-report questionnaire to measure the perceived stress. In 14 items perceived stress is judged by taking into account the previous month's experiences.. Scoring is done using a 5-point Likert scale (0 = never; 4 = very often), with a maximum score (56) representing a higher degree of perceived stress.
Hospital Anxiety and Depression Scale (HADS) | baseline
  Self-report questionnaire of depression and anxiety (14 items) The HADS is aimed at assessing anxiety and depression in a non-psychiatric setting, without questioning physical complaints such as fatigue.The HADS is a self-report questionnaire of 14 items that are answered on the basis of an ordinal scale with four answer options (0-3). Depression and anxiety subscale scores range from 0-21, with higher scores indicating increased depression or anxiety, respectively.
Life Balance Inventory (LBI) | baseline
  LBI is a self-report assessment instrument containing 53 activities and on a dichotomous scale of yes/no, people have to answer, whether or not they do the activity or want to do the activity. For each item scored 'yes', participants have to rate their satisfaction with the amount of time they have spent doing that activity in the past month compared to the amount of time they wanted to do the activity. The possible answers are: "always less than I want (1), sometimes less than I want (2), about right for me (3), sometimes more than I want (2), always more than I want (1)".
  The LBI contains four subscales: (1) Health subscale (ex. Relaxing, getting regular exercise, …), (2) Relationship subscale (ex. Doing things with friends, partner, …), (3) Identity subscale (ex. Taking care of your appearance, participating in religious events, …), (4) Challenge/interest subscale (ex. Working for pay, making music, …).
  Higher scores reflect better life balance.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Kos, PhD, Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - KU Leuven, Department of Rehabilitation Sciences, Leuven
  - National Multiple Sclerosis Center, Melsbroek

IPD SHARING:
Plan to Share IPD: Undecided